CLINICAL TRIAL: NCT01764750
Title: A Prospective Dose-Escalation Trial of the Pharmacokinetics and Preliminary Safety of Intrasite Lyophilized Vancomycin to Prevent Wound Infections in Instrumented Spinal Surgery
Brief Title: Dose Escalation Trial of Intrasite Vancomycin Pharmacokinetics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: awaiting FDA approval for next dose group
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012IntrasiteVanc
Record Dates: First submitted 2012-12-14; First posted 2013-01-10 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Surgical Site Infection
Keywords: Intrasite; Antibiotic; Vancomycin; Infection; Pharmacokinetics
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Dose Intrasite Vancomycin (Experimental): 10 patients will be enrolled to receive low dose (see protocol) intrasite Vancomycin at the time of surgery. This will be the first group enrolled in the dose-escalation trial.
  Interventions: Drug: Intrasite Vancomycin
- Mid-dose Intrasite Vancomycin (Experimental): 10 patients will be enrolled to receive mid-dose intrasite Vancomycin at the time of surgery.
  Interventions: Drug: Intrasite Vancomycin
- High-dose Intrasite Vancomycin (Experimental): 10 patients will be enrolled to receive high-dose intrasite Vancomycin at the time of surgery.
  Interventions: Drug: Intrasite Vancomycin
- Optimally-dosed IV Vancomycin (Active Comparator): 10 patients will be enrolled to receive optimally-dosed IV Vancomycin at the time of surgery and two doses post-operatively (standard peri-operative IV antibiotics)
  Interventions: Drug: IV Vancomycin

INTERVENTIONS:
Drug: Intrasite Vancomycin — Intrasite Vancomycin is placement of lyophilized Vancomycin powder directly into the surgical site at the completion of surgery.
  Arms: High-dose Intrasite Vancomycin; Low Dose Intrasite Vancomycin; Mid-dose Intrasite Vancomycin
Drug: IV Vancomycin — IV Vancomycin is the standard route for systemic antibiotic surgical site wound infection prophylaxis.
  Arms: Optimally-dosed IV Vancomycin

SUMMARY:
Surgical wound infections remain a serious problem despite aseptic techniques and the use of prophylactic systemic antibiotics. Such infections can occur at rates up to ~20% in high-risk patients receiving long segment instrumented spinal fusions for deformity correction and present potentially catastrophic consequences. Given this, the high cost of treatment, and a payer system unable to support such expenses, investigators must make every effort to find new cost-effective ways to prevent these complications.

Increasingly surgeons have sought to address this problem by placing lyophilized Vancomycin into spinal surgery wounds immediately prior to wound closure. This method, known as "intrasite" application, is adapted from techniques used to prevent infection in joint replacement surgeries. The motivation for this practice is to maximize antibiotic concentration within the wound while minimizing systemic concentration and toxicity, (the inverse of the situation when using IV antibiotics). While the popularity of intrasite delivery has grown rapidly, this has occurred without prospective scientific evidence. Recently, three retrospective papers including nearly 2,500 treated patients, indicated that intrasite Vancomycin reduces wound infections without increasing adverse events[1-3]. However, there are no published data on the dosing or pharmacokinetics of intrasite Vancomycin, let alone prospective trials of its efficacy and safety.

The investigators propose to perform the first prospective trial of intrasite Vancomycin pharmacokinetics and safety. Study objectives will include standardizing application and dosing, defining peak/trough concentrations and clearance parameters, verifying bactericidal potency, and dose selection for use in future studies. This will be accomplished by enrolling groups of patients (n=10) to receive one of three doses of intrasite lyophilized Vancomycin (3, 6 or 12 mg/cm2), prior to wound closure. Vancomycin concentrations in venous blood and wound seroma fluid will be measured at regular intervals after surgery to establish pharmacokinetic parameters. Preliminary data regarding local and systemic adverse events including wound healing, fusion rate, and toxicity will be prospectively collected. The ultimate goal of this learning-phase study is to gather sufficient information regarding application, dosing, pharmacokinetics, measurement strategies, and adverse events to prepare for a Phase III efficacy trial.

DETAILED DESCRIPTION:
Despite extremely close attention to aseptic technique and the use of prophylactic IV antibiotics, wound infection rates for posterior instrumented spinal surgery have been as high as ~20% in published studies[4-13]. Such infections can be devastating for patients, frequently requiring multiple re-operations to remove and then replace spinal implants, lengthy hospital stays, prolonged courses of intravenous antibiotics, pain, immobility, and increased risk of other complications. While the cost of the initial surgical episode can be upwards of $250,000, the total cost of care can increase to more than quadruple this number when complications like wound infection occur[14, 15]. Given the impetus to decrease healthcare costs and a federal reimbursement policy denying payment for any care surrounding a wound infection, it is critical to search for cost-effective ways of preventing surgical wound infections[14, 16].

For several decades the standard of care in North America for surgical wound infection prophylaxis has been IV cephalosporin administration within one hour of incision, followed by interval IV dosing for 24 to 48hrs post-procedure[5, 13]. In some settings these antibiotics now effectively treat less than half of identified infection-causing organisms[17, 18]. In response, some groups of surgeons, including at the investigators' own institution, have begun placing lyophilized Vancomycin into the surgical wound bed at the conclusion of the procedure in an effort to further reduce wound infection rates[1-3]. The rationale behind this intrasite antibiotic application is to increase local concentrations of antibiotic to many times the minimally inhibitory concentration (MIC) for even moderately-resistant gram-positive organisms, thereby increasing the bacterial kill rate[3]. It is also thought that local antibiotic application should minimize blood concentrations of the drug, thereby minimizing systemic complications like renal toxicity. Additionally, it is hypothesized that intrasite antibiotic therapy could be less inclined to generate resistant organisms due to a steep concentration gradient from the wound to the systemic circulation. The site of potential infection (the wound) receives a dose of antibiotic vastly exceeding the saturation concentration for bactericidal effect while the systemic concentration remains extremely low. Bacteria should therefore be completely exterminated in the area of the wound or elsewhere exposed to such a minimal concentration of Vancomycin that selection for resistant organisms is avoided.

While none of these hypotheses have been rigorously or prospectively tested, three retrospective studies have recently published a total of 2,479 spinal fusion patients treated with intrasite Vancomycin for wound infection prophylaxis[1-3]. The largest of these studies demonstrated a 0.99% infection rate in the treatment group, among the lowest rates ever published[1]. Two of the studies showed large and statistically significant decreases in the wound infection rate, compared to historical controls, when using intrasite Vancomycin in addition to standard of care IV cephalosporins. Preliminary evidence in one study also indicated high levels of Vancomycin within the wound and low or undetectable levels within the blood following surgery[3]. All of these studies specifically cited that no adverse events had been observed related to the treatment[1-3].

If intrasite Vancomycin proves to be safe and effective for preventing spinal fusion surgical site infections, the treatment will offer great clinical value both for reducing morbidity and also for decreasing large unsupported costs. A future large prospective efficacy trial would be required to provide high-level evidence for this new mode of antibiotic therapy in order to justify wide-spread adoption of the practice in spine surgery. Such data in any population might also be generalizable to surgical wounds at large and prompt a paradigm shift in infection prophylaxis for all types of surgical wounds. The proposed study addresses necessary prerequisites for such a large-scale efficacy trial, including basic pharmacokinetic and preliminary prospective safety data.

ELIGIBILITY:
Inclusion Criteria:

1. Posterior instrumented spinal surgery patients 18 years of age and older with instrumented fusion of at least three vertebral levels

   1. Revision, elderly, obese, and diabetic patients will not be excluded since these patients are known to be at higher risk of wound infection and represent an important fraction of the elective surgical patient population.
2. Patients requiring IV Vancomycin for infection prophylaxis (i.e. due to cephalosporin allergy) will be eligible for participation in the IV Vancomycin group.

Exclusion Criteria:

Intrasite Vancomycin Study Arm Exclusion Criteria

1. Children under 18 years old
2. Patients not receiving instrumentation or having less than three segment surgery

   - therefore having small wound bed surface areas, close operative quarters, and lower infection risk.
3. Patients not receiving wound drains

   * drains provide the conduit for seroma fluid collection
4. Patients with known or suspected current infection
5. Use of systemic or topical antibiotics within 72 hours prior to surgery

   * other than standard pre-op dose of ancef
6. Use of drugs or medications known to significantly increase the risk of renal toxicity within the perioperative period.
7. Patients with known significant allergy to Vancomycin

   - Redman Syndrome patients will not be excluded
8. Use of IV Vancomycin for perioperative infection prophylaxis (for example, in cases of penicillin/cephalosporin allergy) will exclude patients from participation in the intrasite Vancomycin groups of the study.

   * IV Vancomycin Study Arm Exclusion Criteria

<!-- -->

1. Children under 18 years old
2. Patients not receiving instrumentation or having less than three segment surgery - therefore having small wound bed surface areas, close operative quarters, and lower infection risk.
3. Patients not receiving wound drains

   - drains provide the conduit for seroma fluid collection
4. Patients with known or suspected current infection
5. Use of systemic or topical antibiotics within 72 hours prior to surgery

   * other than study related IV Vancomycin
6. Use of drugs or medications known to significantly increase the risk of renal toxicity within the perioperative period.
7. Patients with known significant allergy to Vancomycin

   * Redman Syndrome patients will not be excluded
8. Use of intrasite Vancomycin for infection prophylaxis will exclude patients from participation in the IV Vancomycin study group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Blood Vancomycin Concentration | Post-operatively at daily intervals until surgical drain is removed (average of 4 days after surgery)
  Blood Vancomycin concentration will be measured within two hours post-operatively as well as each morning (between 07:00 and 09:00) until the surgical drain is removed (normally around 4 days after surgery).
Seroma Vancomycin Concentration | Post-operatively at daily intervals until surgical drain is removed (average of 4 days after surgery)
  Seroma Vancomycin concentration will be measured within two hours post-operatively as well as each morning (between 07:00 and 09:00) until the surgical drain is removed (normally around 4 days after surgery).

SECONDARY OUTCOMES:
Blood creatinine concentration | Post-operatively at daily intervals until surgical drain is removed (average of 4 days after surgery)
  Blood serum creatinine concentration will be measured at daily intervals each morning (between 07:00 to 09:00) post-operatively until surgical drain is removed approximately 4 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence F Holekamp, MD, PhD, Principal Investigator — Washington University School of Medicine; Lawrence G Lenke, MD, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Background] Molinari RW, Khera OA, Molinari WJ 3rd. Prophylactic intraoperative powdered vancomycin and postoperative deep spinal wound infection: 1,512 consecutive surgical cases over a 6-year period. Eur Spine J. 2012 Jun;21 Suppl 4(Suppl 4):S476-82. doi: 10.1007/s00586-011-2104-z. Epub 2011 Dec 8. PMID 22160172
- [Background] O'Neill KR, Smith JG, Abtahi AM, Archer KR, Spengler DM, McGirt MJ, Devin CJ. Reduced surgical site infections in patients undergoing posterior spinal stabilization of traumatic injuries using vancomycin powder. Spine J. 2011 Jul;11(7):641-6. doi: 10.1016/j.spinee.2011.04.025. Epub 2011 May 19. PMID 21600853
- [Background] Sweet FA, Roh M, Sliva C. Intrawound application of vancomycin for prophylaxis in instrumented thoracolumbar fusions: efficacy, drug levels, and patient outcomes. Spine (Phila Pa 1976). 2011 Nov 15;36(24):2084-8. doi: 10.1097/BRS.0b013e3181ff2cb1. PMID 21304438
- [Background] Friedman ND, Sexton DJ, Connelly SM, Kaye KS. Risk factors for surgical site infection complicating laminectomy. Infect Control Hosp Epidemiol. 2007 Sep;28(9):1060-5. doi: 10.1086/519864. Epub 2007 Jun 28. PMID 17932827
- [Background] Olsen MA, Nepple JJ, Riew KD, Lenke LG, Bridwell KH, Mayfield J, Fraser VJ. Risk factors for surgical site infection following orthopaedic spinal operations. J Bone Joint Surg Am. 2008 Jan;90(1):62-9. doi: 10.2106/JBJS.F.01515. PMID 18171958
- [Background] Linam WM, Margolis PA, Staat MA, Britto MT, Hornung R, Cassedy A, Connelly BL. Risk factors associated with surgical site infection after pediatric posterior spinal fusion procedure. Infect Control Hosp Epidemiol. 2009 Feb;30(2):109-16. doi: 10.1086/593952. PMID 19125680
- [Background] Pull ter Gunne AF, Cohen DB. Incidence, prevalence, and analysis of risk factors for surgical site infection following adult spinal surgery. Spine (Phila Pa 1976). 2009 Jun 1;34(13):1422-8. doi: 10.1097/BRS.0b013e3181a03013. PMID 19478664
- [Background] Pull ter Gunne AF, Mohamed AS, Skolasky RL, van Laarhoven CJ, Cohen DB. The presentation, incidence, etiology, and treatment of surgical site infections after spinal surgery. Spine (Phila Pa 1976). 2010 Jun 1;35(13):1323-8. doi: 10.1097/BRS.0b013e3181bcde61. PMID 20150831
- [Background] Schimmel JJ, Horsting PP, de Kleuver M, Wonders G, van Limbeek J. Risk factors for deep surgical site infections after spinal fusion. Eur Spine J. 2010 Oct;19(10):1711-9. doi: 10.1007/s00586-010-1421-y. Epub 2010 May 6. PMID 20445999
- [Background] Gerometta A, Rodriguez Olaverri JC, Bitan F. Infections in spinal instrumentation. Int Orthop. 2012 Feb;36(2):457-64. doi: 10.1007/s00264-011-1426-0. Epub 2012 Jan 5. PMID 22218913
- [Background] Li Y, Glotzbecker M, Hedequist D. Surgical site infection after pediatric spinal deformity surgery. Curr Rev Musculoskelet Med. 2012;5(2):111-9. doi: 10.1007/s12178-012-9111-5. Epub 2012 Feb 9. PMID 22315161
- [Background] Pull ter Gunne AF, Hosman AJ, Cohen DB, Schuetz M, Habil D, van Laarhoven CJ, van Middendorp JJ. A methodological systematic review on surgical site infections following spinal surgery: part 1: risk factors. Spine (Phila Pa 1976). 2012 Nov 15;37(24):2017-33. doi: 10.1097/BRS.0b013e31825bfca8. PMID 22565388
- [Background] van Middendorp JJ, Pull ter Gunne AF, Schuetz M, Habil D, Cohen DB, Hosman AJ, van Laarhoven CJ. A methodological systematic review on surgical site infections following spinal surgery: part 2: prophylactic treatments. Spine (Phila Pa 1976). 2012 Nov 15;37(24):2034-45. doi: 10.1097/BRS.0b013e31825f6652. PMID 22648023
- [Background] Graf K, Ott E, Vonberg RP, Kuehn C, Schilling T, Haverich A, Chaberny IF. Surgical site infections--economic consequences for the health care system. Langenbecks Arch Surg. 2011 Apr;396(4):453-9. doi: 10.1007/s00423-011-0772-0. Epub 2011 Mar 15. PMID 21404004
- [Background] Calderone RR, Garland DE, Capen DA, Oster H. Cost of medical care for postoperative spinal infections. Orthop Clin North Am. 1996 Jan;27(1):171-82. PMID 8539047
- [Background] Centers for Medicare and Medicaid Services (CMS), HHS. Medicaid program; payment adjustment for provider-preventable conditions including health care-acquired conditions. Final rule. Fed Regist. 2011 Jun 6;76(108):32816-38. PMID 21644388
- [Background] Klevens RM, Edwards JR, Richards CL Jr, Horan TC, Gaynes RP, Pollock DA, Cardo DM. Estimating health care-associated infections and deaths in U.S. hospitals, 2002. Public Health Rep. 2007 Mar-Apr;122(2):160-6. doi: 10.1177/003335490712200205. PMID 17357358
- [Background] Klevens RM, Morrison MA, Nadle J, Petit S, Gershman K, Ray S, Harrison LH, Lynfield R, Dumyati G, Townes JM, Craig AS, Zell ER, Fosheim GE, McDougal LK, Carey RB, Fridkin SK; Active Bacterial Core surveillance (ABCs) MRSA Investigators. Invasive methicillin-resistant Staphylococcus aureus infections in the United States. JAMA. 2007 Oct 17;298(15):1763-71. doi: 10.1001/jama.298.15.1763. PMID 17940231
- [Background] Mahmood I, Duan J. Population pharmacokinetics with a very small sample size. Drug Metabol Drug Interact. 2009;24(2-4):259-74. doi: 10.1515/dmdi.2009.24.2-4.259. PMID 20408503
- [Background] Lodise TP, Drusano GL, Butterfield JM, Scoville J, Gotfried M, Rodvold KA. Penetration of vancomycin into epithelial lining fluid in healthy volunteers. Antimicrob Agents Chemother. 2011 Dec;55(12):5507-11. doi: 10.1128/AAC.00712-11. Epub 2011 Sep 12. PMID 21911567
- [Background] Rybak MJ. The pharmacokinetic and pharmacodynamic properties of vancomycin. Clin Infect Dis. 2006 Jan 1;42 Suppl 1:S35-9. doi: 10.1086/491712. PMID 16323118
- [Background] Rybak M, Lomaestro B, Rotschafer JC, Moellering R Jr, Craig W, Billeter M, Dalovisio JR, Levine DP. Therapeutic monitoring of vancomycin in adult patients: a consensus review of the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2009 Jan 1;66(1):82-98. doi: 10.2146/ajhp080434. No abstract available. PMID 19106348